CLINICAL TRIAL: NCT00363571
Title: The Effect of Glyceryl Trinitrate (GTN) and Diamox on Cerebral Haemodynamics Judged With the Help of 3-Tesla MRI.
Brief Title: The Effect of Glyceryl Trinitate and Diamox on Cerebral Haemodynamics.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: KA-20060084
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Acetazolamide

INTERVENTIONS:
Drug: GTN, Diamox

SUMMARY:
After infusion / injection of Glyceryl trinitrate and Diamox it is wished to study the effect of drugs on the cerebral haemodynamics such as Cerebral blod flow and cerebral blod volume.

DETAILED DESCRIPTION:
Experimental headache model open a unike opportunity to study the pathophysiological mechanisms behind headache in general and migrane in particular. Previous studies have used various techniques to study the cerebral haemodynamics as a basis for the headache pathophysiology. We wish to use a 3-Tesa MRI so study the cerebral haemodynamics after application of various pharmacological substances.

The most used experimental headache model is the glyceryl trinitrate model (GTN). Where infusion of the NO donor GTN induces headache and changes in the cerebral arteries. On the other hand injection of Diamox (Acetazolamide) apparently causes increase of the cerebral blod flow with out dilation of the arteries. We wish to study the precise effect of GTN and diamox on the cerebral haemodynamics such as Cerebral blod flow (CBF) and Cerebral blod volume (CBV) via a 3-Tesla MRI.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers; men and women age 18-50 years.
* weight 50-100 kg

Exclusion Criteria:

* Tension type headache more then once per month during the last year.
* Other primary headache types.
* Daily use of medication.
* Pregnant or lactating women.
* Headache on the trail day or 24 hours prior to the trial.
* Contraindications to MRI.
* Hypotension og hypertension.
* Other significant medical conditions judged by the doctor in charge.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2006-08; Study Completion 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD,Ph.D, Study Chair — Danish Headache Center
Locations (1):
- Danish Headache Center, Neurological Dep. Glostrup hospital, Glostrup Municipality, Denmark